CLINICAL TRIAL: NCT01002651
Title: In Vivo Evaluation of the Physiological Effects of Arabinoxylan-oligosaccharides (AXOS) in Healthy Subjects: a Randomized, Placebo-controlled, Double-blind, Cross-over Study
Brief Title: In Vivo Evaluation of the Physiological Effects of Arabinoxylan-oligosaccharides (AXOS) in Healthy Subjects (Adults)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fugeia NV (Industry)
Responsible Party: Kristin Verbeke, Ph.D., Katholieke Universiteit Leuven
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ML5282
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: gastrointestinal health; healthy subjects
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Wheat Bran Extract (high dose) (Experimental)
  Interventions: Dietary Supplement: wheat bran extract
- Wheat Bran Extract (low dose) (Experimental)
  Interventions: Dietary Supplement: wheat bran extract
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: wheat bran extract — soft drink comprising high WBE dose and natural flavor and coloring agent, ingestion after breakfast and after dinner
  Other Names: arabinoxylan-oligosaccharides (AXOS)
  Arms: Wheat Bran Extract (high dose); Wheat Bran Extract (low dose)
Dietary Supplement: placebo — soft drink with natural flavor and coloring agent, without WBE, ingestion after breakfast and after dinner
  Arms: placebo

SUMMARY:
The investigational study product used in this clinical trial is a soft drink containing an arabinoxylan-oligosaccharides (AXOS) preparation extracted from wheat bran (hereafter called Wheat Bran Extract, WBE).

The objective of this study is to analyze the effect of the intake of two WBE doses on various parameters of gastrointestinal health. Additionally, safety was analyzed using treatment emergent Adverse Events (AEs) and clinical blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-90 years of age, inclusive
* Regular eating habits
* Body Mass Index (BMI) between 18.5 and 30 kg/m2
* Consent to take in the study product according to the study protocol
* Subject is willing to maintain his or her habitual food and beverage intake throughout the study period (with the exception of omission of prebiotic and probiotic food products as indicated in the study protocol)
* For female volunteers of childbearing potential: not planning to become pregnant during the clinical trial and willing to commit to the use of a medically approved form of contraception

Exclusion Criteria:

* Low-calorie diet or other extreme dietary habits in the 6 weeks before the start of the clinical trial
* Recent use of antibiotics
* Abdominal surgery in the past
* Serious illness within 3 months of start of clinical trial
* Use of medication or dietary supplements known to influence GI tract within two weeks of start of clinical trial. Examples of such medication/dietary supplements are antispasmodics, anti diarrhea medication and/or probiotic medication
* Complete anesthetics within 1 month of the start of the clinical trial
* Chronic GI conditions such as inflammatory bowel disease (IBD), inflammatory bowel syndrome (IBS), chronic constipation, history of frequent diarrhea, clinically important lactose intolerance
* Allergy for wheat products
* Celiac disease
* For female volunteers: pregnant or lactating
* Alcohol abuse
* Smoking more than 5 cigarettes per day
* Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the subject at undue risk.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Bifidobacteria content in feces | day 19 or 20 of each intervention
butyric acid content in feces | day 19 or 20 of each intervention
p-cresol content in urine | day 19-21 of each intervention
stool frequency | third week of each intervention

SECONDARY OUTCOMES:
adverse events | whole study
clinical blood parameters | day 21 of each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Willem Broekaert, Ph.D., Study Director — Fugeia NV
Locations (1):
- Department of Gastrointestinal Research, Laboratory Digestion and Absorption, Leuven, Belgium